CLINICAL TRIAL: NCT04169412
Title: Resuscitation Failure, Protein Carbonyl and Receptor Interacting Protein Kinase 3 as Mortality Predictor in Septic Patient
Brief Title: Resuscitation Failure, Oxidative Stress, and Necroptosis as Mortality Predictor in Septic Patient
Status: Completed | Type: Observational
Sponsor: Universitas Sriwijaya (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Mayang Indah Lestari, Principal Investigator, Universitas Sriwijaya
Other Study IDs: 047/kepkrsmhfkunsri/2019
Record Dates: First submitted 2019-11-17; First posted 2019-11-19 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Resuscitation Failure, High PCO Level, High RIPK3 Level: 1. Resuscitation failure was defined as lactate level ≥2 mmol/L or lactate reduction <20% hour-4 after initial sepsis recognition.
  2. High PCO level was defined as PCO level ≥ cut off point.
  3. High RIPK3 level was defined as PCO level ≥ cut off point.
  Interventions: Diagnostic Test: Blood Collection
- Resuscitation Success, Low PCO Level, Low RIPK3 Level: 1. Resuscitation success was defined as lactate level <2 mmol/L or lactate reduction ≥20% hour-4 after initial sepsis recognition.
  2. Low PCO level was defined as PCO level < cut off point.
  3. Low RIPK3 level was defined as PCO level < cut off point.
  Interventions: Diagnostic Test: Blood Collection

INTERVENTIONS:
Diagnostic Test: Blood Collection — Blood Gas Analysis using Stat Profile pHOx® Series (nova biomedical, Waltham, U.S.) and Enzym-linked Immunosorbent Assay (ELISA) using Bio-Rad (Bio-Rad Laboratories, California, U.S.)

SUMMARY:
Resuscitation failure, oxidative stress and necroptosis were able to predict mortality in septic patient

DETAILED DESCRIPTION:
This prospective cohort study was conducted at resuscitation room and ICU of Mohammad Hoesin hospital, a single tertiary teaching hospital in Palembang, South Sumatera. This study was started after ethical and location authorization were unleashed in February to August 2019. Inclusion criteria were patients aged 18 years old or above who met Sepsis-3 definition and diagnosed with sepsis. Exclusion criteria were patients whose family did not give any consent to participate, not treated at the ICU, had a late diagnosis (>24 h), pregnant, and diagnosed with brain dead. Drop out criteria including patients who died <4 h after diagnosed and could not be followed in 28 days. Investigators were trained to identified all eligible subjects. All the subjects had a standard resuscitation and their blood was taken to be examined at the laboratory. Subjects were observed in 28 days whether there were any mortality or not. Failed resuscitation defined by examined lactate level ≥ 2 mmol/L or lactate reduction <20%. Data was statistically analyzed with STATA™

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years old or above
* Diagnosed sepsis using Sepsis-3 definition

Exclusion Criteria:

* Participants whose family did not give any consent to participate
* Not treated at the ICU
* Had a late diagnosis (>24 h)
* Pregnant
* Brain dead

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Resuscitation room and ICU
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
The Ability of Resuscitation Failure, Protein Carbonyl (PCO) and Receptor Interacting Protein Kinase 3 (RIPK3) for Predicting Mortality in Septic Patients | 28 days
  Probability of Mortality in Septic Patients with Resuscitation Failure, High PCO Level and High RIPK3 Level

SECONDARY OUTCOMES:
How Sensitive and Specific Protein Carbonyl (PCO) Level for Predicting Mortality in Septic Patients? | 28 days
  Sensitivity and Specificity of PCO Level for Predicting Mortality in Septic Patients
How Sensitive and Specific Receptor Interacting Protein Kinase 3 (RIPK3) Level for Predicting Mortality in Septic Patients? | 28 days
  Sensitivity and Specificity of RIPK3 Level for Predicting Mortality in Septic Patients

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Hoesin Central General Hospital, Palembang, South Sumatera, Indonesia

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Rhee C, Dantes R, Epstein L, Murphy DJ, Seymour CW, Iwashyna TJ, Kadri SS, Angus DC, Danner RL, Fiore AE, Jernigan JA, Martin GS, Septimus E, Warren DK, Karcz A, Chan C, Menchaca JT, Wang R, Gruber S, Klompas M; CDC Prevention Epicenter Program. Incidence and Trends of Sepsis in US Hospitals Using Clinical vs Claims Data, 2009-2014. JAMA. 2017 Oct 3;318(13):1241-1249. doi: 10.1001/jama.2017.13836. PMID 28903154
- [Background] Dantes RB, Epstein L. Combatting Sepsis: A Public Health Perspective. Clin Infect Dis. 2018 Sep 28;67(8):1300-1302. doi: 10.1093/cid/ciy342. PMID 29846544
- [Background] Marshall JC, Vincent JL, Guyatt G, Angus DC, Abraham E, Bernard G, Bombardier C, Calandra T, Jorgensen HS, Sylvester R, Boers M. Outcome measures for clinical research in sepsis: a report of the 2nd Cambridge Colloquium of the International Sepsis Forum. Crit Care Med. 2005 Aug;33(8):1708-16. doi: 10.1097/01.ccm.0000174478.70338.03. PMID 16096445
- [Background] Weiss SL, Deutschman CS. Elevated malondialdehyde levels in sepsis - something to 'stress' about? Crit Care. 2014 Mar 19;18(2):125. doi: 10.1186/cc13786. PMID 25029036
- [Background] Weinlich R, Oberst A, Beere HM, Green DR. Necroptosis in development, inflammation and disease. Nat Rev Mol Cell Biol. 2017 Feb;18(2):127-136. doi: 10.1038/nrm.2016.149. Epub 2016 Dec 21. PMID 27999438
- [Background] Duprez L, Takahashi N, Van Hauwermeiren F, Vandendriessche B, Goossens V, Vanden Berghe T, Declercq W, Libert C, Cauwels A, Vandenabeele P. RIP kinase-dependent necrosis drives lethal systemic inflammatory response syndrome. Immunity. 2011 Dec 23;35(6):908-18. doi: 10.1016/j.immuni.2011.09.020. PMID 22195746
- [Result] Levy B. Lactate and shock state: the metabolic view. Curr Opin Crit Care. 2006 Aug;12(4):315-21. doi: 10.1097/01.ccx.0000235208.77450.15. PMID 16810041
- [Result] Jansen TC, van Bommel J, Schoonderbeek FJ, Sleeswijk Visser SJ, van der Klooster JM, Lima AP, Willemsen SP, Bakker J; LACTATE study group. Early lactate-guided therapy in intensive care unit patients: a multicenter, open-label, randomized controlled trial. Am J Respir Crit Care Med. 2010 Sep 15;182(6):752-61. doi: 10.1164/rccm.200912-1918OC. Epub 2010 May 12. PMID 20463176
- [Result] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283
- [Result] Yu B, Tian HY, Hu ZJ, Zhao C, Liu LX, Zhang Y, Zhu GJ, Wang LT, Wu XH, Li J. [Comparison of the effect of fluid resuscitation as guided either by lactate clearance rate or by central venous oxygen saturation in patients with sepsis]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2013 Oct;25(10):578-83. doi: 10.3760/cma.j.issn.2095-4352.2013.10.002. Chinese. PMID 24119693
- [Result] Mahmoodpoor A, Shadvar K, Saghaleini SH, Koleini E, Hamishehkar H, Ostadi Z, Nader ND. Which one is a better predictor of ICU mortality in septic patients? Comparison between serial serum lactate concentrations and its removal rate. J Crit Care. 2018 Apr;44:51-56. doi: 10.1016/j.jcrc.2017.10.019. Epub 2017 Oct 17. PMID 29065350
- [Result] Mantzarlis K, Tsolaki V, Zakynthinos E. Role of Oxidative Stress and Mitochondrial Dysfunction in Sepsis and Potential Therapies. Oxid Med Cell Longev. 2017;2017:5985209. doi: 10.1155/2017/5985209. Epub 2017 Aug 20. PMID 28904739
- [Result] Galley HF. Oxidative stress and mitochondrial dysfunction in sepsis. Br J Anaesth. 2011 Jul;107(1):57-64. doi: 10.1093/bja/aer093. Epub 2011 May 19. PMID 21596843
- [Result] Costa NA, Gut AL, Azevedo PS, Tanni SE, Cunha NB, Fernandes AAH, Polegato BF, Zornoff LAM, de Paiva SAR, Balbi AL, Ponce D, Minicucci MF. Protein carbonyl concentration as a biomarker for development and mortality in sepsis-induced acute kidney injury. Biosci Rep. 2018 Jan 25;38(1):BSR20171238. doi: 10.1042/BSR20171238. Print 2018 Feb 28. PMID 29263144
- [Result] He S, Huang S, Shen Z. Biomarkers for the detection of necroptosis. Cell Mol Life Sci. 2016 Jun;73(11-12):2177-81. doi: 10.1007/s00018-016-2192-3. Epub 2016 Apr 11. PMID 27066893
- [Result] Wang B, Li J, Gao HM, Xing YH, Lin Z, Li HJ, Wang YQ. Necroptosis regulated proteins expression is an early prognostic biomarker in patient with sepsis: a prospective observational study. Oncotarget. 2017 Sep 20;8(48):84066-84073. doi: 10.18632/oncotarget.21099. eCollection 2017 Oct 13. PMID 29137405
- [Result] Casserly B, Phillips GS, Schorr C, Dellinger RP, Townsend SR, Osborn TM, Reinhart K, Selvakumar N, Levy MM. Lactate measurements in sepsis-induced tissue hypoperfusion: results from the Surviving Sepsis Campaign database. Crit Care Med. 2015 Mar;43(3):567-73. doi: 10.1097/CCM.0000000000000742. PMID 25479113
- [Result] Levy MM, Evans LE, Rhodes A. The Surviving Sepsis Campaign Bundle: 2018 update. Intensive Care Med. 2018 Jun;44(6):925-928. doi: 10.1007/s00134-018-5085-0. Epub 2018 Apr 19. No abstract available. PMID 29675566
- [Result] Lokhandwala S, Andersen LW, Nair S, Patel P, Cocchi MN, Donnino MW. Absolute lactate value vs relative reduction as a predictor of mortality in severe sepsis and septic shock. J Crit Care. 2017 Feb;37:179-184. doi: 10.1016/j.jcrc.2016.09.023. Epub 2016 Oct 6. PMID 27771598
- [Result] Barreiro E. Role of Protein Carbonylation in Skeletal Muscle Mass Loss Associated with Chronic Conditions. Proteomes. 2016 May 6;4(2):18. doi: 10.3390/proteomes4020018. PMID 28248228
- [Result] Dalle-Donne I, Giustarini D, Colombo R, Rossi R, Milzani A. Protein carbonylation in human diseases. Trends Mol Med. 2003 Apr;9(4):169-76. doi: 10.1016/s1471-4914(03)00031-5. PMID 12727143
- [Result] Dalle-Donne I, Rossi R, Giustarini D, Milzani A, Colombo R. Protein carbonyl groups as biomarkers of oxidative stress. Clin Chim Acta. 2003 Mar;329(1-2):23-38. doi: 10.1016/s0009-8981(03)00003-2. PMID 12589963
- [Result] Suzuki YJ, Carini M, Butterfield DA. Protein carbonylation. Antioxid Redox Signal. 2010 Mar;12(3):323-5. doi: 10.1089/ars.2009.2887. No abstract available. PMID 19743917
- [Result] Abu-Zidan FM, Plank LD, Windsor JA. Proteolysis in severe sepsis is related to oxidation of plasma protein. Eur J Surg. 2002;168(2):119-23. doi: 10.1080/11024150252884359. PMID 12113269
- [Result] Andresen M, Regueira T, Bruhn A, Perez D, Strobel P, Dougnac A, Marshall G, Leighton F. Lipoperoxidation and protein oxidative damage exhibit different kinetics during septic shock. Mediators Inflamm. 2008;2008:168652. doi: 10.1155/2008/168652. PMID 18566692
- [Result] Costa NA, Gut AL, Azevedo PS, Fernandes AAH, Polegato BF, Cunha NB, Bachiega TF, Lourenco MAM, Junior ELF, Zornoff LAM, de Paiva SAR, Minicucci MF. Protein Carbonyl, But Not Malondialdehyde, Is Associated With ICU Mortality in Patients With Septic Shock. J Intensive Care Med. 2019 Aug;34(8):669-673. doi: 10.1177/0885066617710218. Epub 2017 May 19. PMID 28521594
- [Result] Dhuriya YK, Sharma D. Necroptosis: a regulated inflammatory mode of cell death. J Neuroinflammation. 2018 Jul 6;15(1):199. doi: 10.1186/s12974-018-1235-0. PMID 29980212
- [Result] Ma KC, Schenck EJ, Siempos II, Cloonan SM, Finkelsztein EJ, Pabon MA, Oromendia C, Ballman KV, Baron RM, Fredenburgh LE, Higuera A, Lee JY, Chung CR, Jeon K, Yang JH, Howrylak JA, Huh JW, Suh GY, Choi AM. Circulating RIPK3 levels are associated with mortality and organ failure during critical illness. JCI Insight. 2018 Jul 12;3(13):e99692. doi: 10.1172/jci.insight.99692. PMID 29997296